CLINICAL TRIAL: NCT01017042
Title: Open-Label Pharmacokinetic Study of a Low-Dose Acute Gout Regimen
Brief Title: Pharmacokinetic Study of an Acute Gout Regimen
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mutual Pharmaceutical Company, Inc. (Industry)
Responsible Party: Vice President, Branded Products and Medical Affairs, Mutual Pharmaceutical Company, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MPC-004-07-1003
Record Dates: First submitted 2009-08-12; First posted 2009-11-20 (Estimated); Results first posted 2009-11-20 (Estimated); Last update posted 2009-11-20 (Estimated); Status verified 2009-10

CONDITIONS: Pharmacokinetics
Keywords: healthy; blood levels
MeSH Terms: interventions — Colchicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- colchicine (Experimental): colchicine 1.2mg by mouth initially then an additional 0.6mg orally 1 hour later (1.8mg over 2 hours)
  Interventions: Drug: colchicine tablets

INTERVENTIONS:
Drug: colchicine tablets — colchicine 1.2mg initially; then an additional 0.6mg orally 1 hour later (1.8mg over 2 hours)
  Other Names: COLCRYS TM

SUMMARY:
This study aims to characterize the pharmacokinetic profile of colchicine after a regimen of 1.8 mg over two hours. A secondary goal is to evaluate the safety and tolerability of this regimen in healthy volunteers. To this end, all study subjects will be monitored for adverse effects throughout the entire study period.

DETAILED DESCRIPTION:
This study aims to characterize the pharmacokinetic profile of colchicine and its three main metabolites, after a regimen of 1.8 mg over two hours. After a fast of at least 10 hours, fifteen healthy non-smoking, non-obese, non-pregnant adult volunteers between the ages of 18 and 55 will be given colchicine 1.2 mg (2 x 0.6 mg) orally followed by an additional single 0.6mg dose one hour later. Fasting will continue for 4 hours after the first dose at which time a standardized meal will be served. Blood will be drawn from all participants at times sufficient to adequately define the pharmacokinetics of colchicine and its 3 major metabolites, 2, 3 and 10 demethylcolchicine. A further goal of this study is to evaluate the safety and tolerability of this regimen in healthy volunteers. To this end, subjects will be monitored throughout participation in the study for adverse reactions to the study drug and/or procedures. Seated and standing blood pressure and pulse will be measured prior to the first dose and 0.5, 1, 2, 4, and 12 hours post-dose. Twelve-lead electrocardiograms will be obtained at the same time points. All adverse events whether elicited by query, spontaneously reported, or observed by clinic staff will be evaluated by the Investigator and reported in the subject's case report form.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18-55 years of age, non smoking and non-pregnant (postmenopausal, surgically sterile or using effective contraceptive measures) weighing at least 55kg and within 15% of ideal body weight.

Exclusion Criteria:

* Recent participation (within 30 days) in other research studies
* Recent significant blood donation
* Pregnant or lactating
* Test positive at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), or hepatitis C virus (HCV)
* Recent (2-year) history or evidence of alcoholism or drug abuse
* History or presence of significant cardiovascular, pulmonary, hepatic, renal, haematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease
* Subjects who have used any drugs or substances known to inhibit or induce cytochrome (CYP) P450 enzymes and/or P-glycoprotein (P-gp) within 30 days prior to the first dose and throughout the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2007-09; Primary Completion 2007-09 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony R Godfrey, Pharm.D., Principal Investigator — PRACS Institiute, Ltd.
Locations (1):
- PRACS Institute, Ltd. - Cetero Research, Fargo, North Dakota, United States

REFERENCES:
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html
- See also: Daily Med - Posting of Recently Submitted Labeling to the FDA — http://dailymed.nlm.nih.gov/dailymed/about.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Oral Colchicine 1.2mg + 0.6mg: On the morning of day one after a fast of at least 10 hours, all study participants received colchicine 1.2mg by mouth initially then an additional 0.6mg orally 1 hour later (1.8mg over 2 hours) Blood was drawn at times sufficient to characterize the pharmacokinetics of Colchicine under this therapeutic regimen.
Period: Overall Study
Arm/Group | Oral Colchicine 1.2mg + 0.6mg
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Oral Colchicine 1.2mg + 0.6mg
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 28.9 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration
Description: The maximum or peak concentration that the drug reaches in the plasma.
Time Frame: Pharmacokinetic samples collected pre-dose and 0.5, 1 hour (prior to the second dose), and 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, and 48 hours post-dose (relative to the first dose) and 72 and 96 hours post-dose (on an outpatient basis).
Measure: Mean (Standard Deviation); unit: picograms/ml
Arm/Group | Oral Colchicine 1.2mg + 0.6mg
Number analyzed (Participants) | 13
picograms/ml | 6192.77 (2433.7)

2. Secondary Outcome: Electrocardiogram Corrected QT Interval (QTcF)
Description: Corrected QT interval by Fridericia's formula -Measured at baseline, 0.5, 1, 2, and 4 hours
Time Frame: Measured at baseline, 0.5, 1, 2, and 4 hours
Population: All participants
Measure: Mean (Standard Deviation); unit: Milliseconds
Groups:
- Corrected QTc Interval (Baseline): colchicine 1.2mg by mouth initially then an additional 0.6mg orally 1 hour later (1.8mg over 2 hours) QTc corrected by Fridericia's formula (Baseline)
- Corrected QTc Interval (0.5 Hour): colchicine 1.2mg by mouth initially then an additional 0.6mg orally 1 hour later (1.8mg over 2 hours) QTc corrected by Fridericia's formula (0.5hour)
- Corrected QTc Interval (1 Hour): colchicine 1.2mg by mouth initially then an additional 0.6mg orally 1 hour later (1.8mg over 2 hours) QTc corrected by Fridericia's formula (1 hour)
- Corrected QTc Interval (2 Hour): colchicine 1.2mg by mouth initially then an additional 0.6mg orally 1 hour later (1.8mg over 2 hours) QTc corrected by Fridericia's formula (2 hour)
- Corrected QTc Interval (4 Hour): colchicine 1.2mg by mouth initially then an additional 0.6mg orally 1 hour later (1.8mg over 2 hours) QTc corrected by Fridericia's formula (4 hour)
Arm/Group | Corrected QTc Interval (Baseline) | Corrected QTc Interval (0.5 Hour) | Corrected QTc Interval (1 Hour) | Corrected QTc Interval (2 Hour) | Corrected QTc Interval (4 Hour)
Number analyzed (Participants) | 13 | 13 | 13 | 13 | 13
Milliseconds | 402.28 (19.66) | 397.38 (18.37) | 399.26 (20.59) | 401.51 (20.64) | 402.38 (23.16)

3. Primary Outcome: Area Under the Concentration Time Curve From Time Zero to the Time of Last Measured Concentration (96 Hours) (AUC 0-t)
Description: The area under the plasma concentration versus time curve beginning from the first dose until the last quantifiable concentration (96hours), calculated by the linear trapezoidal rule.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg-hr/ml
Arm/Group | Oral Colchicine 1.2mg + 0.6mg
Number analyzed (Participants) | 13
pg-hr/ml | 43787.55 (11437.48)

4. Primary Outcome: Area Under The Concentration Time Curve From Zero Through Infinity (AUC∞)
Description: The area under the plasma concentration versus time curve extrapolated to infinity.
  AUC∞ is calculated as the sum of Total AUC0-t plus the ratio of the last measurable plasma concentration to the elimination rate constant
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg-hr/ml
Arm/Group | Oral Colchicine 1.2mg + 0.6mg
Number analyzed (Participants) | 13
pg-hr/ml | 52070.06 (13689.27)

ADVERSE EVENTS:
Arm/Group | Oral Colchicine 1.2mg + 0.6mg
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 5
OTHER ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Oral Colchicine 1.2mg + 0.6mg
Abdominal Pain , Upper (Gastrointestinal disorders) | 1/13 (1)
Diarrhea (Gastrointestinal disorders) | 2/13 (2)
Dyspepsia (Gastrointestinal disorders) | 1/13 (1)
Nausea (Gastrointestinal disorders) | 1/13 (1)
Headache (Nervous system disorders) | 2/13 (2)
Hot Flush (Vascular disorders) | 1/13 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days